CLINICAL TRIAL: NCT06727162
Title: The Value of Contrast-enhanced Ultrasound in Assessing the Response of Cervical Lymph Nodes After Neoadjuvant Chemoimmunotherapy for Head and Neck Squamous Cell Carcinoma
Brief Title: The Value of CEUS in Assessing the Response of Cervical Lymph Nodes After NACI for HNSCC
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-873-01
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Contrast-Enhanced Ultrasound — Participants are scanned in a supine position with the neck fully exposed. A routine ultrasound examination is first performed to assess the cervical lymph nodes. Assessment includes: number, size, location (zones I-VII), structure, echogenicity, margin, shape, hilum, calcification, and vascular distribution.
  After the routine ultrasound scan, the ultrasound system is switched to dual contrast-enhanced ultrasound mode. Sonazoid (GE Healthcare) is then administered intravenously through the antecubital vein at a dose of 0.015 mL/kg, followed by an injection of 5 mL of physiological saline. A timer is started after the injection, and video recording is made during the vascular phase from 5 to 60 seconds.

SUMMARY:
The head and neck squamous cell carcinoma is the sixth most common malignant tumor worldwide. For patients with locally advanced head and neck cancer, neoadjuvant therapy is recommended before surgery, including neoadjuvant chemotherapy and immunotherapy. There is a significant variation in patients' responses to neoadjuvant therapy, with approximately 37%-52% of patients achieving a complete pathological response after neoadjuvant therapy. Current research mainly focuses on the efficacy evaluation of the primary tumor, while there is less research on the treatment efficacy evaluation of cervical lymph nodes. In clinical practice, accurate assessment of the status of cervical lymph nodes after neoadjuvant chemoimmunotherapy in patients with squamous cell carcinoma of the head and neck can directly affect the choice of treatment plan by clinicians, reducing unnecessary neck dissection. In recent years, contrast-enhanced ultrasound has been widely used in the diagnosis of thyroid cancer and other head and neck tumors, as well as in the assessment of the benign and malignant nature of cervical lymph nodes. This study aims to explore the value of contrast-enhanced ultrasound in the assessment of cervical lymph nodes after neoadjuvant chemoimmunotherapy in squamous cell carcinoma of the head and neck, in order to guide clinicians in formulating personalized treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* (1) Histopathologically confirmed head and neck squamous cell carcinoma; (2) Received neoadjuvant chemoimmunotherapy; (3) Diagnosed with cN+ by CT/MRI before treatment; (4) Underwent radical surgical treatment plus cervical lymph node dissection at this center.

Exclusion Criteria:

* (1) Did not receive a full course of neoadjuvant therapy; (2) History of treatment for head and neck; (3) Clinical evidence of distant metastasis found during preoperative examination.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with HNSCC, who treated in Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | From enrollment to the end of surgery at 10 weeks
  Sensitivity = True Positives / (True Positives + False Negatives).
Specificity | From enrollment to the end of surgery at 10 weeks
  Specificity = True Negatives / (True Negatives + False Positives).
Positive Predictive Value | From enrollment to the end of surgery at 10 weeks
  Positive Predictive Value = True Positives / (True Positives + False Positives)
Negative Predictive Value | From enrollment to the end of surgery at 10 weeks
  Negative Predictive Value = True Negatives / (True Negatives + False Negatives)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China